CLINICAL TRIAL: NCT03989674
Title: Glycaemic Index (GI) Evaluation of Carbohydrate-based Food with Functional Ingredients Derived from Food Sources
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Collaborators: National University Health System, Singapore (Other)
Responsible Party: Principal Investigator, Mei Hui Liu, Senior Lecturer, National University of Singapore
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: H-17-064
Record Dates: First submitted 2019-06-14; First posted 2019-06-18 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2021-07

CONDITIONS: Postprandial Hyperglycemia
Keywords: Glycemic index; Postprandial hyperglycemia; Anthocyanin; Black rice
MeSH Terms: conditions — Hyperglycemia | interventions — Anthocyanins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- White bread (No Intervention)
- Anthocyanin-fortified bread (2% w/w) (Experimental)
  Interventions: Dietary Supplement: Anthocyanin
- Anthocyanin-fortified bread (4% w/w) (Experimental)
  Interventions: Dietary Supplement: Anthocyanin

INTERVENTIONS:
Dietary Supplement: Anthocyanin — 25% w/w anthocyanin extract obtained from black rice
  Arms: Anthocyanin-fortified bread (2% w/w); Anthocyanin-fortified bread (4% w/w)

SUMMARY:
In Singapore, the Ministry of Health has declared a "War on Diabetes" and major efforts will be made to develop and deploy programs to prevent diabetes. One of the cornerstones of diabetes management involves dietary modifications to reduce postprandial hyperglycaemia. However, implementation of a low GI diet is highly complex requiring the individual to choose foods from a long list which are primarily based on western consumption patterns. Many foods in the Asian diet, which largely consist of carbohydrates such as white rice, noodles and other flour based products, are not represented. An alternative solution will require innovative ways to alter commonly available food products that will not only help reduce postprandial glycaemia but also preserve the sensory characteristics of the foods to create a new generation of food products both functional and palatable. One such approach is the incorporation of plant compounds that lower the glucose absorption from foods. The aim of the project is to measure the GI of carbohydrate-based food with edible plant derived molecules. Natural, plant-derived anthocyanin will be incorporated into bread to produce low GI bread. Anthocyanins are well known for its anti-oxidant activity and recent studies reported that anthocyanins also had an inhibitory activity against digestive enzymes that break down carbohydrates. It can potentially inhibit amylase, and suppress the increase in postprandial glucose level from starch. Bread is a carbohydrate-rich product, which contains a high amount of rapidly digestible starch, and therefore many of them have a high GI. This study aims to determine the glycaemic effects of anthocyanin fortified bread. The effort is designed to enable and inform population interventions that will have an impact on the health of the population in a sustainable manner by introducing innovative foods into the food supply that are 'health promoting' based on rigorous human experiments and are acceptable to the public and other major stakeholders.

ELIGIBILITY:
Inclusion Criteria:

* Ability to give informed consent
* Age between 21-65 years old
* Overtly healthy males or females, as determined by medical history, physical examination and laboratory results within normal reference range for the population or investigator site, or results with acceptable deviations that are judged to be not clinically significant by the investigator
* Males and females with stable medical problems that, in the investigator's opinion, will not significantly alter the performance of the biomarker panel, will not place the subject at increased risk by participating in the study, and will not interfere with interpretation of the data.
* Not on any regular medications (western / traditional medicine). Nutritional supplements with established chemical composition that can be ascertained and clearly recorded is acceptable.

However, subjects using traditional medicine (with compositions that cannot be ascertained) will be excluded in this study.

* Have venous access sufficient to allow for blood sampling as per the protocol
* Reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures (participants are required to fast overnight for 10-12h before each visit).

Exclusion Criteria:

* History or presence of current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, malignancy or neurological disorders capable of significantly altering the performance of the biomarker panel; or of interfering with the interpretation of data
* Known or ongoing psychiatric disorders within 3 years
* Regularly use known drugs of abuse within 3 years
* Women who are pregnant or lactating
* Have donated blood of more than 500 mL within 4 weeks of study enrolment
* Have an average weekly alcohol intake that exceeds 21 units per week (males) and 14 units per week (females):

  * 1 unit = 12 oz or 360 mL of beer;
  * 5 oz or 150 mL of wine;
  * 1.5 oz or 45 mL of distilled spirits
* Uncontrolled hypertension (blood pressure [BP] >160/100mmHg
* Active infection requiring systemic antiviral or antimicrobial therapy that will not be completed prior to Study Day 1
* Treatment with any investigational drug, or biological agent within one (1) month of screening or plans to enter into an investigational drug/ biological agent study during the duration of this study
* Known allergy to insulin
* History of bleeding diathesis or coagulopathy
* Any of the following laboratory values at screening:

Fasting glucose >=126mg/dL(>=7mmol/L) or 2 hour post-prandial glucose >=200mg/dL (>=11.1mmol/L)

* Clinically significant (as determined by investigator) abnormalities on laboratory examination that will increase risk to the patient or interfere with data integrity
* Have any other conditions, which, in the opinion of the Investigator would make the subject unsuitable for inclusion, or could interfere with the subject participating in or completing the study
* Significant change in weight (+/- 5%) during the past month

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-10-27 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Glycemic index | 2 hours
  Change in incremental area-under-curve (min*mmol/L)

SECONDARY OUTCOMES:
Anthocyanin and metabolite bioavailability | 0 minutes, 60 minutes, 120 minutes
  Change in anthocyanin and anthocyanin metabolite concentrations (mg/L)
Oxidative stress | 0 minutes, 60 minutes, 120 minutes
  Change in total F2-isoprostane concentration (mg/L)

CONTACTS AND LOCATIONS:
Overall Officials: Mei Hui Liu, PhD, Principal Investigator — National University of Singapore
Locations (1):
- Investigational Medicine Unit, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sui X, Zhang Y, Zhou W. Bread fortified with anthocyanin-rich extract from black rice as nutraceutical sources: Its quality attributes and in vitro digestibility. Food Chem. 2016 Apr 1;196:910-6. doi: 10.1016/j.foodchem.2015.09.113. Epub 2015 Oct 9. PMID 26593572
- [Background] van Dam RM, Naidoo N, Landberg R. Dietary flavonoids and the development of type 2 diabetes and cardiovascular diseases: review of recent findings. Curr Opin Lipidol. 2013 Feb;24(1):25-33. doi: 10.1097/MOL.0b013e32835bcdff. PMID 23254472
- [Background] Zhang PW, Chen FX, Li D, Ling WH, Guo HH. A CONSORT-compliant, randomized, double-blind, placebo-controlled pilot trial of purified anthocyanin in patients with nonalcoholic fatty liver disease. Medicine (Baltimore). 2015 May;94(20):e758. doi: 10.1097/MD.0000000000000758. PMID 25997043